CLINICAL TRIAL: NCT05057455
Title: Effectiveness of the Cytokine Hemadsorption on the Clinical Progression and Mortality of Intensive Care Patients With Sepsis
Brief Title: Effectiveness of the Cytokine Hemadsorption on Sepsis
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, IKUPELI, investigator, Biruni University
Other Study IDs: BIRUNI 2
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Interleukin-6

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients diagnosed with sepsis or septic shock: compare the laboratory and clinical results of cytokine hemadsorption as an immunomodulation therapy in ICU patients diagnosed with sepsis or septic shock.
  Interventions: Procedure: cytokine hemadsorption

INTERVENTIONS:
Procedure: cytokine hemadsorption — the laboratory and clinical results of cytokine hemadsorption as an immunomodulation therapy in ICU patients diagnosed with sepsis or septic shock.

SUMMARY:
In this prospective study, we aimed to compare the laboratory and clinical results of cytokine hemadsorption as an immunomodulation therapy in ICU patients diagnosed with sepsis or septic shock.

ELIGIBILITY:
Inclusion Criteria:

* the patients were the available data of clinical and laboratory diagnosis of sepsis and septic shock
* detection of gram-negative bacterial agent in blood or sputum culture.
* patients who had the shock symptoms such as hypotension, tachycardia or fever during the course of sepsis.

Exclusion Criteria:

* had uncontrolled hemorrhage,
* diagnosed with cardiac failure at stage 4 or renal failure at stage 4 or hepatic liver failure at stage 4
* cancer at the end stage or admitted with acute coronary syndrome.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this one-centered study, we prospectively analyzed the outcomes and laboratory findings of 39 patients diagnosed with sepsis from 01 Jan 2020 to 30 December 2020 hospitalized in ICU.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
IL-6 | 1 YEARS
  levels of IL-6

CONTACTS AND LOCATIONS:
Locations (1):
- Ilke Kupeli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bahar I, Oksuz H, Senoglu N, Demirkiran H, Aydogan M, Tomak Y, Comez M, Bayrakci S, Gonullu E, Berktas M. Compliance With the Surviving Sepsis Campaign Bundle: A Multicenter Study From Turkey. Cureus. 2021 May 12;13(5):e14989. doi: 10.7759/cureus.14989. PMID 34131534
- [Result] Houschyar KS, Pyles MN, Rein S, Nietzschmann I, Duscher D, Maan ZN, Weissenberg K, Philipps HM, Strauss C, Reichelt B, Siemers F. Continuous hemoadsorption with a cytokine adsorber during sepsis - a review of the literature. Int J Artif Organs. 2017 May 29;40(5):205-211. doi: 10.5301/ijao.5000591. Epub 2017 May 19. PMID 28525674
- [Result] Ye Q, Wang B, Mao J. The pathogenesis and treatment of the ;Cytokine Storm' in COVID-19. J Infect. 2020 Jun;80(6):607-613. doi: 10.1016/j.jinf.2020.03.037. Epub 2020 Apr 10. PMID 32283152
- [Result] Bonavia A, Groff A, Karamchandani K, Singbartl K. Clinical Utility of Extracorporeal Cytokine Hemoadsorption Therapy: A Literature Review. Blood Purif. 2018;46(4):337-349. doi: 10.1159/000492379. Epub 2018 Sep 3. PMID 30176653